CLINICAL TRIAL: NCT04635085
Title: The Feasibility and Preliminary Effects of an Empowerment-based Cognitive Behavioural Therapy for Insomnia on Sleep, Cognitive Function and Health--related Quality of Life in Persons With Mild Cognitive Impairment
Brief Title: A Mixed Method Pilot Study for Patients With Mild Cognitive Impairment and Insomnia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Polly Wai-Chi Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HKWC-2020-0029
Record Dates: First submitted 2020-11-05; First posted 2020-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment; Insomnia
Keywords: mild cognitive impairment; Empowerment; insomnia; sleep; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowerment-based Cognitive behavioral therapy for insomnia for MCI (intervention) (Experimental): Participants in the intervention group will participate in a 12-week empowerment-based CBT-I comprising face-to-face sessions supplemented with telephone follow-ups.
  Interventions: Behavioral: Empowerment-based Cognitive behavioral therapy for insomnia for MCI
- Social Activities provided by the community centers (active control) (No Intervention): The control group will not receive any structured cognitive training or sleep promoting interventions during the study period. The participants in the control group will continue to participate in the social activities offered by the elderly community centers. They have access to the newspapers, board games and computer facility in the centers. Upon completion of collecting all evaluation data for both groups at the three different time points, the empowerment-based CBT-I will be offered to participants in the control group.

INTERVENTIONS:
Behavioral: Empowerment-based Cognitive behavioral therapy for insomnia for MCI — Participants in the intervention group will participate in a 12-week empowerment-based CBT-I comprising face-to-face sessions supplemented with telephone follow-ups. In total, six face-to-face sessions (90 minutes/session) will be conducted in a small group format with 6-8 participants in a group.
  Arms: Empowerment-based Cognitive behavioral therapy for insomnia for MCI (intervention)

SUMMARY:
Dementia is irreversible, incurable and devastating. It is thus imperative to preserve cognition at the pre-dementia stage. Mild cognitive impairment (MCI) refers to the reversible intermediate clinical state between normal age-related cognitive decline and dementia. Because no pharmacological treatments have proved to be effective, risk factor modification remains the cornerstone in preventing progression from MCI to dementia. Insomnia is an emerging risk factor now being associated with cognitive decline, and it affects up to 59% of persons with MCI. Compelling evidence shows that sleep is vital for memory consolidation, and it mediates the deposition of amyloid-β and tau proteins in the brain. Despite these findings, minimal research has done to evaluate sleep-promoting interventions on the cognitive function of persons with MCI. Non-pharmacological interventions remain the treatment of choice for managing insomnia, particularly the older population. These interventions require individuals to actively participate in the treatment process. Yet, the cognitive impairment and neuropsychiatric symptoms in persons with MCI create challenges for them. An empowerment approach with interactive teaching strategies and experiential learning may be the best method of engaging people in the learning process and arousing their inherent capacity to maintain behavioral modifications. This study aims to examine the feasibility and preliminary effects of an empowerment-based cognitive behavioral therapy for insomnia (CBT-I) in persons with MCI and sleep problems. The researchers will compare the effects of this intervention by comparing with the standard care.

DETAILED DESCRIPTION:
The proposed study will have two aims: i) to determine the feasibility of an empowerment-based CBT-I in MCI persons; and ii) to examine the preliminary effects of the empowerment-based CBT-I on sleep, cognitive outcomes and HRQoL in persons with MCI

Study design This is a mixed-method study with a single-blinded parallel-group randomized controlled trial (RCT) and a qualitative study to determine the feasibility and preliminary effects of the empowerment-based CBT-I on sleep, cognitive outcomes and HRQoL in persons with MCI. Eligible participants will be recruited from the elderly community centers operated by two non-governmental organizations in Hong Kong. After collecting the baseline data (T0), participants will be randomly assigned into the intervention group and control group with block randomization to ensure even distribution of participants in the two study groups over the study period. A computer-generated random sequence will be used to determine the block size (6, 8 and 10) and respective study group allocation in a 1:1 ratio. To ensure allocation concealment, the group allocation will be determined according to the random sequence codes placed in sealed opaque envelopes. Participants in the intervention group will receive the empowerment-based CBT-I, whereas the control group will receive usual care provided by the community centers. A total of 60 participants (i.e., 30/study arm) will be recruited for this pilot RCT. Upon completion of the RCT, ten participants in the intervention group will be invited to have an individual qualitative interview to gather their in-depth comments about the feasibility and acceptability of the empowerment-based CBT-T intervention. The collected information will be used to optimize the procedures and process of the future main study. To reduce contamination of the control group, the intervention sessions will be delivered in a private room of the study sites. The participants in the intervention group will be advised not to share the content with other members in the centers. Nonetheless, the active ingredients of the intervention are the intensive interactions between the intervener and the participants, which is less likely to be replicated and disclosed by the participants.

Study Interventions Intervention group: Empowerment-based CBT-I for MCI Participants in the intervention group will participate in a 12-week empowerment-based CBT-I comprising face-to-face sessions supplemented with telephone follow-ups. In total, six face-to-face sessions (90 minutes/session) will be conducted in a small group format with 6-8 participants in a group and two 30-minute individual sessions will be scheduled over eight weeks, with the individual sessions arranged in the 4th and 7th week, and this is then followed by two bi-weekly telephone follow-ups. The face-to-face sessions will cover the following core areas in CBT-I: i) sleep education, ii) sleep hygiene and relaxation, iii) sleep restriction, iv) stimulus control and v) cognitive therapy. The first five sessions will cover these core areas, and a booster session will then follow to summarize the key components of CBT-I and equip the participants with relapse-prevention strategies when sleeping problems recur. The content of the CBT-I components complies with the recommendations for managing chronic insomnia by major international sleep associations.

A five-step empowerment approach will be adopted to implement each face-to-face session to facilitate goal attainment and behavioral maintenance. At the beginning of each session, the intervener will encourage the participants to discuss their usual practice or beliefs about sleep or insomnia related to the core area of that week, then deliver a structured educational session about the topic area. The rationales and explicit methods of how to carry out the suggested behaviors will be stated. The content will emphasize assisting participants to understand the linkage between their usual practice (behaviors/thoughts) and the consequences to sleep disruption. The intervener will then facilitate the participants to identify the discrepancies between their usual practice/dysfunctional beliefs and the recommended best practice for sleep improvement/beliefs that favor better sleep. Easy-to-understand comic stories will be incorporated to illustrate the more abstract concepts about dysfunctional beliefs related to insomnia (for the session on cognitive therapy) and bed-sleep association (for the session on stimulus control). The intervener will also highlight the possible consequences of these discrepancies on brain health. The intervener will then assist participants to set self-directed goals related to these areas. During this process, the intervener will work collaboratively with the participants and ensure that the goals are achievable yet challenging. The intervener will also work with the participants to develop an action plan for achieving the goals set during each session. After action-planning, a subsequent interactive skill-building session will ensure that participants acquire the skills required to perform specific behaviors. A scenario-based approach will be adopted to train the participants on how to maintain the recommended behaviors. The intervener will make use of group dynamics by encouraging the discussion among the peers of successful actions, feelings, concerns and perceived barriers to goal achievement. Various memory compensatory strategies will be used to reinforce the educational content, such as memory aids (e.g., memory notebooks, calendars and to-do lists) and mnemonic strategies. Each subsequent session will begin with a discussion of progress in goal attainment and challenges and barriers encountered while implementing the action plan set during the preceding week.

The intervener will provide continuous support through individualized one-to-one face-to-face meetings (7th and 9th week) and telephone calls (three bi-weekly calls on 8th, 10th and 12th week) upon the completion of all the group-based sessions. A personal record containing the participants' demographic and clinical profile, endorsed dysfunctional beliefs and attitudes about sleep, self-directed goals and action plans will be created to facilitate the individualized face-to-face sessions and telephone support. The intervener will monitor participants' adherence to the recommended behaviors and goal attainment progress, identify barriers in real-life settings and provide methods of resolving them. The advice and counseling given will be documented to guide subsequent telephone calls.

Control group: Usual care The control group will not receive any structured cognitive training or sleep promoting interventions during the study period. The participants in the control group will continue to participate in the social activities offered by the elderly community centers. They have access to the newspapers, board games and computer facility in the centers.

ELIGIBILITY:
Inclusion Criteria:

* aged >=50 years
* living in the community
* Independence in daily living as evaluated through the clinical interview
* Presence of cognitive complaints, defined as >= 3 complaints on the Memory Inventory for Chinese
* Abnormal objective cognitive performance defined as <-1.5 standard deviations from age
* Education-matched normal persons on the Montreal Cognitive Assessment Hong Kong Version (HK-MoCA)
* Persons with poor sleep quality that can be assessed by the Pittsburgh Sleep Quality Index, with a global PSQI score of >5

Exclusion Criteria:

* Persons with confirmed dementia
* Persons with known psychiatric conditions
* Persons with impaired communication
* Persons with sleep disorders with an organic cause (e.g., sleep apnea, or restless legs syndrome) or due to a medical problem (e.g., pain)
* Persons with the use of hypnotics and other medications known to affect sleep (e.g., steroids, anxiolytics)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Sleep on the 19 item The Pittsburgh Sleep Quality (PSQI) Index at the 12th week and 3 months | Change from Baseline Chinese PSQI at the 12th week (after the intervention) and 3 months (follow up)]
  The Chinese PSQI is a validated, self-reported instrument for assessing sleep disturbance over the month. A 3-point Likert scale is used to each item (0=no difficulty; to 3 =severe difficulty). Possible total score ranging from 0-21. MCI persons with global score>5 will be eligible for inclusion.
Changes from Baseline in Insomnia Severity on the 7-item The Chinese version of the Insomnia Severity Index (ISI-C)at the 12th week and 3 months | Change from Baseline ISI-C at the 12th week (after the intervention) and 3 months (follow up)]
  The ISI-C is a validated, self-reported instrument for assessing the perceived insomnia severity, consequences of insomnia and the degree of distress related to insomnia. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), Possible a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
An Actiwatch, which contains an accelerometer (during sleep for a consecutive seven-day period) | Change from Baseline the frequency of body movement at the 12th week (after the intervention) and 3 months (follow up)]
  to record the frequency of body movement, will be used to objectively assess sleep patterns automatically.
An Actiwatch, which contains an accelerometer (during sleep for a consecutive seven-day period) | Change from Baseline the intensity of body movement at the 12th week (after the intervention) and 3 months (follow up)]
  to record the intensity of body movement, will be used to objectively assess sleep patterns automatically.
An Actiwatch, which contains an accelerometer (during sleep for a consecutive seven-day period) | Change from Baseline sleep parameters at the 12th week (after the intervention) and 3 months (follow up)]
  To record the sleep parameters include total sleep time (TST), sleep latency (SL), wake after sleep onset (WASO) and the ratio of total sleep time (TST) to sleep efficiency (SE) of sleep, will be used to objectively assess sleep patterns automatically.
Changes from the Cantonese version of the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | Change from Baseline ADAS-Cog at the 12th week (after the intervention) and 3 months (follow up)]
  The ADAS-Cog is a validated instrument for assessing language, memory in order to detect the subtle cognitive changes. The standard ADAS-cog includes the following 11 items, with a possible Total scoring range of 0 - 70. The ADAS score is based on the number of errors made in each item. A score of 70 represents the most severe impairment and 0 represents the least impairment.
Changes from the Hong Kong List Learning Test (HKLLT) | Change from Baseline HKLLT at the 12th week (after the intervention) and 3 months (follow up)]
  The HKLLT is a validated instrument for assessing complex attention, executive function and task switching. Participants were required to learn a list of 16 Chinese words through three learning trials. After 10 and 30 min delay, they were asked to recall as many words as possible. The total number of recalled words after a delay was used to reflect verbal memory ability. A low score on Trial 1, with normal performance on Trial 3 and total learning, is considered to reflect problems in auditory attention spam, but intact learning ability. Poor scores on all three learning trials provide evidence for acquisition problems in learning and memory. The T-score range from <20 to >/= 65. The score of >=65 represents superior and <20 represents the severely impaired.
the Color Trail Test (CCT) | Change from Baseline the CCT at the 12th week (after the intervention) and 3 months (follow up)]
  CCT is a validated instrument for assessing complex attention, executive function and task switching. Time taken to complete each part of the CTT is recorded in seconds and is compared to normative data. Qualitative aspects of the performance that may be indicative of brain dysfunction (e.g. near misses, prompts required, sequencing errors for color and number) are also recorded. The CTT manual reports that it takes 3-8 minutes to complete the CTT. A task is discontinued if the client takes longer than 240 seconds to complete it. Performance time <60 seconds on the CTT was found to predict passing the on-road evaluation, whereas >60 seconds was predictive of failing
The Chinese Hong Kong version of the Short Form Health Survey (SF-12) | Change from Baseline SF-12 at the 12th week (after the intervention) and 3 months (follow up)]
  SF-12 is a validated instrument for assessing the general health of people, both physical and mental well-being. A mental component score and a physical component score are reported as Z-scores (different compared to the population average, 12 are both 50 points). The standard deviation is 10 points, so each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Polly, Wai Chi LI, Principal Investigator — The School of Nursing, The University of Hong Kong
Locations (1):
- Polly Wai Chi, Hong Kong, Please Select, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li PWC, Yu DSF, Wong CWY. An empowerment-based cognitive behavioural therapy for persons with mild cognitive impairment and insomnia: Protocol for a mixed-method pilot study. J Adv Nurs. 2021 Apr;77(4):2054-2063. doi: 10.1111/jan.14740. Epub 2021 Jan 13. PMID 33438783

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04635085/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04635085/ICF_000.pdf